CLINICAL TRIAL: NCT03462303
Title: Modulation of Cognitive Flexibility by Tyrosine Depletion and Transcranial Direct Current Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: SheffieldHallamAquili2018
Record Dates: First submitted 2018-02-20; First posted 2018-03-12 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Cognitive Flexibility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- tDCS sham + balanced drink (Placebo Comparator)
  Interventions: Combination Product: Sham tDCS and balanced drink
- tDCS sham + tyrosine depleted drink (Experimental)
  Interventions: Combination Product: Sham tDCS and tyrosine depleted drink
- tDCS anodal + balanced drink (Experimental)
  Interventions: Combination Product: Anodal tDCS and balanced drink
- tDCS anodal +tyrosine depleted drink (Experimental)
  Interventions: Combination Product: Anodal tDCS and tyrosine depleted drink

INTERVENTIONS:
Combination Product: Sham tDCS and tyrosine depleted drink — Transcranial direct current stimulation (sham) of the dlPFC in combination with a tyrosine and phenylalanine free product.
  Arms: tDCS sham + tyrosine depleted drink
Combination Product: Anodal tDCS and tyrosine depleted drink — Transcranial direct current stimulation (anodal) of the dlPFC in combination with a tyrosine and phenylalanine free product.
  Arms: tDCS anodal +tyrosine depleted drink
Combination Product: Sham tDCS and balanced drink — Transcranial direct current stimulation (sham) of the dlPFC in combination with a drink containing both tyrosine and phenylalanine.
  Arms: tDCS sham + balanced drink
Combination Product: Anodal tDCS and balanced drink — Transcranial direct current stimulation (anodal) of the dlPFC in combination with a drink containing both tyrosine and phenylalanine.
  Arms: tDCS anodal + balanced drink

SUMMARY:
The dorsolateral prefrontal cortex (dlPFC) and dopamine (DA) have been implicated in the control of cognitive flexibility. However, while a great deal of what it is know regarding a causative relationship between cognitive flexibility and its neuronal underpinning comes from animal studies, human data have largely been correlational (i.e. imaging investigations). In a recent study, the current research group examined whether putative increases in dopamine levels through tyrosine administration and blockage of these by cathodal (i.e. inhibitory) transcranial direct current stimulation (tDCS) of the dlPFC could be causally related to cognitive flexibility as measured by task switching and reversal learning.

The next step involves finding a way of lowering dopamine concentrations while anodal (i.e. excitatory) stimulation of the dlPFC is applied and cognitive flexibility measured. One experimental approach to reduce global DA synthesis and transmission is through acute phenylalanine and tyrosine depletion (APTD). This dietary intervention involves the administration of an amino-acid mixture lacking in tyrosine and phenylalanine, which can be used to selectively lower DA synthesis in humans.

ELIGIBILITY:
Inclusion Criteria:

* Either male or female
* You are aged between 18 and 30 years
* You are in good health
* You agree to fast overnight prior to testing

Exclusion Criteria:

* Are suffering from cardiac, hepatic, renal, or neurological disorders
* Damaged or diseased skin on your face and scalp, or a sensitive scalp
* A history of alcohol or drug addiction, or severe psychiatric illness
* Are in drug treatment which may lower seizure threshold (i.e. epilepsy)
* You are pregnant
* Slept less than 6 hours prior to coming to the lab
* Suffer from phenylketonuria
* A history of or current experience of migraine or headaches
* A history of or current use of antidepressants
* A history of or current use of tyrosine supplements
* Consume more than five beverages containing caffeine per day

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in cognitive flexibility performance | Measured over 5 hours four times.1st measurement taken at baseline (i.e. time 0). 2nd measurement taken 120 minutes after measurement 1. 3rd measurement taken 220 minutes after measurement 1. 4th measurement taken 270 minutes after measurement 1.
  Measured using Wisconsin Card Sorting Test
Change in cognitive flexibility performance | Measured over 5 hours. 1st measurement taken at baseline (i.e. time 0). 2nd measurement taken 120 minutes after measurement 1. 3rd measurement taken 220 minutes after measurement 1. 4th measurement taken 270 minutes after measurement 1.
  Measured using Probabilistic Reversal Learning

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology labs, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT03462303/SAP_000.pdf